CLINICAL TRIAL: NCT07369323
Title: Erector Spinae Plane Block for Postoperative Pain After Kidney Transplantation: A Prospective Study"
Brief Title: Erector Spinae Plane Block in Kidney Transplant Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Özlem Sezen, assosiate proffesor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 514/250/6
Record Dates: First submitted 2025-05-25; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-05

CONDITIONS: Kidney Failure
Keywords: renal transplantation; erector spine plane block; pain management
MeSH Terms: conditions — Renal Insufficiency; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control group (Other): tandard postoperative analgesia protocol was applied. Intravenous paracetamol (1 g/8 hours) was administered. ESP block not implemented
  Interventions: Other: ESP block

INTERVENTIONS:
Other: ESP block — USG-guided unilateral ESP block at T9 level (0.25% bupivacaine 20 ml)

SUMMARY:
Use of postoperative analgesia in kidney transplant recipients has always been challenging due to several issues: potential nephrotoxicity of nonsteroidal anti- inflammatory drugs and the reduced clearance of morphine metabolites due to transient renal impairment.Moreover, many patients with end-stage renal disease on dialysis are hepatitis C or hepatitis B virus positive, and the use of other effective analgesics, such as acetaminophen, is limited.The use of regional analgesia methods for postoperative analgesia can also be a useful option for more adequate control in these patients. Currently, methods of fascial trunk nerve blocks (including rectus sheath block, different types of transversus abdominis plane block, and erector spinae plane [ESP] block) have been shown to be effective components of multimodal anesthesia in various fields of surgery.In this study, investigators evaluated the effectiveness of ESP block in the postoperative period after kidney transplant.The aim of this prospective, randomized controlled trial is to evaluate the effects of erector spinae plane block on postoperative analgesia quality, opioid consumption, and side effect profile in kidney transplant patients.The study included a total of 40 patients aged 18-65 years with ASA physical status II-III who were scheduled for elective kidney transplantation. All patients received standard general anesthesia. Anesthesia induction was achieved with propofol (2-2.5 mg/kg), fentanyl (1-2 µg/kg), and rocuronium (0.6 mg/kg). Anesthesia maintenance was provided with 6% desflurane and a 50% oxygen-air mixture.ESPB Group: USG-guided unilateral ESP block at T9 level (0.25% bupivacaine 20 ml)

* Control Group: no block applied
* All patients received standard postoperative analgesia protocol. Intravenous paracetamol (1 g/8 hours) was given. Intravenous tramadol (100 mg) was administered as rescue analgesic when VAS ≥ 4.

ELIGIBILITY:
Inclusion Criteria:

* All patients had end-stage renal disease due to chronic glomerulonephritis _ physical status of class 3 on American Society of Anesthesiologists classification.

Exclusion Criteria:

* ASA 4

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Postoperrative VAS scores at 24 hours | postoperative 24 hours
  Postoperative Vas scores at 15 minutes, 1 hour, 2 hours, 6 hours, 12 hours, and 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr Lutfi Kırdar City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No